CLINICAL TRIAL: NCT05589012
Title: Evaluation of Viral Replication by Tonate Virus (TONV) and Zika Virus (ZIKV), Within an ex Vivo Trophoblast and Placental Model
Acronym: ZITOPEx
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01318-31
Record Dates: First submitted 2022-08-22; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-08

CONDITIONS: Zika Virus Infection
Keywords: trophoblast; placenta
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Human placentas and trophoblasts (biological waste) from uncomplicated pregnancies.: The placentas will be collected following a birth by caesarean section after oral and written information by delivery of the information note for women who have had a normal singleton pregnancy at term.
  Similarly, trophoblasts are collected following endo-uterine aspiration in the context of voluntary termination of pregnancy.
  * Cell line and virus
  * Infection of human placental culture explants
  * Determination of viral load in tissues by qRT-PCR
  Interventions: Biological: Cell line and virus; Biological: Infection of human placental culture explants; Biological: Determination of viral load in tissues by qRT-PCR

INTERVENTIONS:
Biological: Cell line and virus — C6/36 cells will be cultured in L15 culture medium (Leibovitz's L-15 medium), supplemented with 5% FBS (Fetal Bovine Serum) and 1% penicillin/streptomycin at 28°C in a humidified atmosphere containing 5% C02. ZIKV and TONV will be expanded and titrated using C6/36 cells. The viral stock will be aliquoted in 100 µL aliquots and stored at -80°C.
Biological: Infection of human placental culture explants — Placental tissues will be handled within one hour of delivery. The chorionic villi will be dissected into 5mm sections and the tissues washed abundantly, minimum 3 times with a standard culture medium (RPMI-1640 supplemented with 10% heat-inactivated fetal calf serum (FCS), 1% L-Glutamine and 1% Penicillin/Streptomycin) to remove maternal blood, membranes and blood clots.
  Collagen gel sponges will be placed in 6-well plate wells containing 3mL of culture medium (RPMI-1640 supplemented with 15% heat-inactivated fetal bovine serum (FCS), 1% Penicillin/streptomycin, 0 1% Gentamycin, 1% Amphotericin B, 1% L-Glutamine, 1% non-essential amino acid, 1% sodium pyruvate) per well. Chorionic villi will be dissected into 5mm sections and placed on top of collagen gel sponges at the interface between culture medium and air.
Biological: Determination of viral load in tissues by qRT-PCR — The tissues will be lysed by mechanical disruption in a lysis buffer + 4%TCEP (Tris(2-carboxyethyl)phosphine hydrochloride) (Machery-Nagel ref: 740395.107) with the Precellys system. The lysed tissues will be diluted in 100 mg/mL of Macherey-Nagel lysis buffer, aliquoted and stored at -80°C until extraction. Total RNA will be extracted in duplicate using the Nucleospin 96 RNA Core kit (Macherey Nagel ref: 740466.4), following the supplier's instructions.
  Standard samples, controls and ZIKV and TONV viral RNA will be extracted and tested in parallel under the same conditions. The extracted RNA will be subjected to reverse transcriptase, using the Superscript One-Step RT-qPCR kit (Invitrogen ref: 11732088) according to the manufacturer's recommendations, with a probe and primer specific for ZIKV and TONV.

SUMMARY:
Prospective, non-interventional study carried out after culturing placental trophoblastic tissue ex vivo and infection with Zika and Tonate

DETAILED DESCRIPTION:
The analysis will relate for each virus studied + control + favipiravir to 1 placenta in the 1st trimester and 1 placenta at term.

2 experiments per virus will be planned.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Singleton pregnancy of normal course, at term, birth by caesarean section OR
* Trophoblast from Voluntary Termination of Pregnancy (IVG), after endo-uterine aspiration

Exclusion Criteria:

* Need for pathological, genetic or bacteriological examination of the placenta
* Multiple pregnancy
* HBV+ (Hepatitis B positive), HCV+ (Hepatitis C positive) , known CMV seroconversion during pregnancy (CytoMégaloVirus)
* Immunosuppression (drugs, corticosteroids, etc.)
* Diabetes
* Pre eclampsia
* Intrauterine growth retardation (IUGR),
* Vascular or placental pathology.
* Refusal to participate
* Patient under guardianship / curatorship / security measure
* Patient under AME (state medical aid)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
To assess the replication potential of TONV and ZIKV after placenta infection ex vivo. | inclusion
  Determine the viral load (RT-qtPCR) of TONV and ZIKV after placenta infection, ex vivo in RNA copies/mL

SECONDARY OUTCOMES:
Validate the ex vivo placental model for TONV. | Inclusion
  Analysis of viral load in placental explants for TONV in RNA copies/mL
Compare viral infection of the placenta at different terms of pregnancy (first trimester and term). | first trimester
  Analysis of the viral load according to the term in RNA copies/mL
Compare viral infection of the placenta at different terms of pregnancy (first trimester and term). | first trimester
  Analysis of gene expression of the different cytokines according to the term in RNA copies/mL
Compare viral infection of the placenta at different terms of pregnancy (first trimester and term). | first trimester
  Analysis of the histological lesions according to the term in RNA copies/mL
Compare viral infection of the placenta at different terms of pregnancy (first trimester and term). | term
  Analysis of the viral load according to the term in RNA copies/mL
Compare the placental infection of TONV versus ZIKV. | inclusion
  Analysis of viral load depending on the virus (ZIKV vs TONV) in RNA copies/mL
Compare the placental infection of TONV versus ZIKV. | inclusion
  Analysis of gene expression of different cytokines depending on the virus (ZIKV vs TONV) in RNA copies/mL
Compare the placental infection of TONV versus ZIKV. | inclusion
  Analysis of histological lesions depending on the virus (ZIKV vs TONV) in RNA copies/mL
Highlight the cellular targets of TONV. | inclusion
  Histological analysis and labeling of TONV cells in RNA copies/mL
Highlight the cellular targets of TONV. | inclusion
  Histological analysis and labeling of placental cells in RNA copies/mL

IPD SHARING:
Plan to Share IPD: No